CLINICAL TRIAL: NCT03840317
Title: Randomized, Parallel-arm, Controlled Trial of Senl_1904A and Senl_1904B Autologous CAR-T Cell Injections in the Treatment of Relapsed and Refractory Acute B Lymphocytic Leukemia(r/r B-ALL)
Brief Title: Senl_1904A and Senl_1904B Chimeric Antigen Receptor （CAR） T-Cell in the Treatment of r/ r Acute B Lymphocytic Leukemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hebei Senlang Biotechnology Inc., Ltd. (Industry)
Collaborators: Hebei Yanda Ludaopei Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Senl_1904A & Senl_1904B CAR-T
Record Dates: First submitted 2019-01-27; First posted 2019-02-15 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Acute Lymphocytic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Senl_1904A CD19 CAR-T (Experimental): Autologous CD19-targeting CAR T cells, dosage 3*10^5/kg, intravenous injection once
  Interventions: Biological: Autologous CD19-targeting CAR T cells
- Senl_1904B CD19 CAR-T (Experimental): Autologous CD19-targeting CAR T cells,dosage 3*10^5/kg, intravenous injection once
  Interventions: Biological: Autologous CD19-targeting CAR T cells

INTERVENTIONS:
Biological: Autologous CD19-targeting CAR T cells — Autologous CD19-targeting CAR T cells

SUMMARY:
This is an open, two arms, mask phase I clinical study to evaluate efficacy and safety of two different chimeric antigen receptor T cell immunotherapies (Senl_1904A and Senl_1904B) targeting cluster of differentiation antigen 19 （CD19） in the treatment of Acute lymphocytic Leukemia. A total of 20 patients are planned to be enrolled following up half a year.

DETAILED DESCRIPTION:
The CARs consist of an anti-CD19 single-chain variable fragment（scFv） that was derived from the FMC63 mouse hybridoma, a portion of the human CD137（4-1BB） molecule, and the intracellular component of the human CD3ζ molecule. Autologous T cells will be gene engineered with the CAR gene using a lentivirus vector. Compared to Senl_1904A, Senl_1904B has a higher and more stable transfection efficiency and secretes lower levels of cytokines in functional assays, thus having the potential to significantly reduce the incidence of serious adverse events while ensuring the same complete response rate. Prior to T cell infusion, the patients will be subjected to preconditioning treatment. After T cell infusion, the patients will be evaluated for one month after infusion for adverse reactions and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with acute lymphocytic leukemia who voluntarily signed informed consent and met the following criteria:

  1. Patients with relapsed and refractory acute B lymphocytic leukemia with any of the following:

     1. Recurrence after remission by chemotherapy or autologous stem cell transplantation (including B-ALL patients with bone marrow recurrence of morphology and recurrence of micro-residual );
     2. Primary B-ALL patients who cannot be completely relieved by repeated chemotherapy twice or more;
     3. High-risk initial onset B-ALL patients not completely relieved after 1 or 2 times of chemotherapy but not suitable for re-chemotherapy ;
  2. Tumor cells confirmed CD19 positive by Flow cytometry (FCM)
  3. For B-ALL patients with simple extramedullary recurrence , there must be at least one evaluable lesion;
  4. Eastern Cooperative Oncology Group (ECOG) ≤ 2 points;
  5. Age 3 - 65 years old;
  6. The bone marrow tumor load value (morphology) > 5% at the time of enrollment;
  7. The main organ function needs to meet the above conditions: cardiac ultrasound or multiple gated image acquisition analysis （MUGA） scan indicate the cardiac ejection fraction is ≥50% , and there is no obvious abnormality in the electrocardiogram; blood oxygen saturation≥90%; creatinine ≤1.6mg/dl; alanine amino transferase (ALT) and Aspartate transaminase (AST)≤3 times normal range, total bilirubin（TBil） ≤2.0mg/dl;
  8. The expected survival time is longer than 3 months;
  9. The pregnancy test for women of childbearing age must be negative; Subjects with a pregnancy plan must agree to take contraception before the enrollment study and after the study lasts for one year; if the subject is pregnant or suspects of pregnancy, the investigator should be notified immediately
  10. An informed consent form is required.

Exclusion Criteria:

* 1) Severe cardiac insufficiency; 2) A history of severe pulmonary dysfunction; 3) Combined with other malignant tumors; 4) Combined with serious infections or persistent infection and cannot be effectively controlled; 5) Combined with metabolic diseases (except DM); 6) Combined with severe autoimmune diseases or congenital immune defects; 7) Active hepatitis (HBV DNA or HCVRNA detection positive); 8) HIV infection or syphilis infection; 9) A history of severe allergies to biological products (including antibiotics); 10) Subjects with recurrence after allogeneic hematopoietic stem cell transplantation 11) chronic lymphocytic leukemia（CLL） /myeloproliferative neoplasms with acute lymphoid transformation or CLL transform to ALL ; 12) Any drug that has been used against graft-versus-host disease（GVHD） for nearly 4 weeks, such as methotrexate or other chemotherapeutic drugs, mycophenolate mofetil, immunosuppressive antibodies, etc.; 13) Subjects who have received any anti-CD19 medication; 14) Subjects who have used anti-cluster of differentiation antigen 20（CD20） drugs (such as rituximab) for nearly 4 weeks; 15) Subjects who have participated in any other clinical drug trials in the past six months; 16) Female patients who are pregnant and lactating, or have a pregnancy plan within 12 months; 17) The investigator believes that it may increase the risk of the subject or interfere with the outcome of the test (with a history of severe mental illness, drug abuse and history of addiction).

Exit criteria：

1. The subjects request to withdraw from the study before CAR-T infusion
2. The subjects seriously violate the protocol
3. Before CAR-T infusion, the following indicators are still abnormal after treatment:

   Platelets <20x10^9/L, hemoglobin ≤80g/L, peripheral finger oxygen <90%, AST / ALT / alkaline phosphatase（ALP） ≥ 2.5 upper limits of normal（ULN）, total bilirubin ≥ 1.5ULN , creatinine clearance rate <70ml / min, left ventricular ejection fraction <50%, the researcher judged that the test needs to be terminated early;
4. The therapeutic dose of steroids was not stopped within 72 hours prior to CAR-T infusion and the investigator determined that the trial needs to be terminated . However, the following physiologically acceptable doses of steroids are permissible: hydrocortisone or equivalent <6-12 mg/m2/day ;
5. Not enough T cells for manufacture standard CAR-T cells
6. Other serious adverse events occurred
7. MRD become negative after preconditioning regiment

Ages: 3 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-01-02 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Tumor load | up to one month
  Tumor load will be quantified with radiology, bone marrow and/or blood samples dependent on diagnosis.

SECONDARY OUTCOMES:
CAR T cell expansion | up to one month
  The percentage of CAR-T cells (CAR+/CD3+ T cells) in the bone marrow samples, quantified by flow cytometry.
CAR T cell persistence | up to one month
  The method to detect CAR-T cell persistence is by determining the exact copies of CAR per ug DNA in BM through quantitative polymerase chain reaction（qPCR）

CONTACTS AND LOCATIONS:
Overall Officials: Peihua Lu, PhD&MD, Principal Investigator — Hebei Yanda Ludaopei Hospital
Locations (1):
- Hebei Yanda Ludaopei Hospital, Langfang, Hebei, China

REFERENCES:
- [Derived] Ho JY, Wang L, Liu Y, Ba M, Yang J, Zhang X, Chen D, Lu P, Li J. Promoter usage regulating the surface density of CAR molecules may modulate the kinetics of CAR-T cells in vivo. Mol Ther Methods Clin Dev. 2021 Mar 13;21:237-246. doi: 10.1016/j.omtm.2021.03.007. eCollection 2021 Jun 11. PMID 33869653